CLINICAL TRIAL: NCT03555825
Title: Burke-Hocoma Efficiency Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Burke Medical Research Institute (Other)
Collaborators: Hocoma (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BRC540
Record Dates: First submitted 2018-05-15; First posted 2018-06-14 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Hemiparesis; Hemiplegia
MeSH Terms: conditions — Paresis; Hemiplegia

STUDY DESIGN:
Intervention Model Description: Group 1: 60 minutes of Armeo treatment, 3 times per week for 6 weeks. (Half the patients will be assigned to 1:1 therapy and the other half to 2:1 therapy) Group 2: 30 minutes of Armeo treatment, 3 times per week for 6 weeks. (Half the patients will be assigned to 1:1 therapy and the other half to 2:1 therapy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- 60 Minutes ArmeoSpring (1:1) (Active Comparator): 60 minutes of therapy 3x per week for 6 weeks working one-on-one with a clinician for duration of session.
  Interventions: Device: Hocoma ArmeoSpring
- 60 Minutes ArmeoSpring (2:1) (Experimental): 60 minutes of therapy 3x per week for 6 weeks with one clinician supervising 2 participants.
  Interventions: Device: Hocoma ArmeoSpring
- 30 Minutes ArmeoSpring (1:1) (Active Comparator): 30 minutes of therapy 3x per week for 6 weeks working one-on-one with a clinician for duration of session.
  Interventions: Device: Hocoma ArmeoSpring
- 30 Minutes ArmeoSpring (2:1) (Experimental): 30 minutes of therapy 3x per week for 6 weeks with one clinician supervising 2 participants.
  Interventions: Device: Hocoma ArmeoSpring

INTERVENTIONS:
Device: Hocoma ArmeoSpring — A spring-loaded upper extremity exoskeleton with 3 joints and 6 degrees of freedom. Participants use the more affected upper extremity to control and engage in therapeutic games.

SUMMARY:
The ArmeoSpring device is an exoskeleton (3 joints and 6 degrees of freedom) with integrated springs. The investigators hypothesize that 3 days of training for 6 weeks with the Hocoma Armeo Spring device will be efficient and more effective than one on one ArmeoSpring therapy.

DETAILED DESCRIPTION:
In the proposed study, 20 stable subacute and chronic stroke patients will be placed in two groups: 2:1 treatment for 3 weeks (2 patients on 2 robots with one therapist; 60 minutes on robot) then 1 on 1 intervention with the therapist (60 minutes of Hocoma Armeo Spring robotic training) or visa versa. Patients will be assessed using robotic kinematics and standardized occupational therapy motor assessments. The extreme precision afforded by robotic physical rehabilitation therapies makes them an appealing and growing field in rehabilitation.

Determining efficiency of new technologies, while maintaining the highest quality of care, is of priority in the medical field at this time. Devices such as the ArmeoSpring could lead to reduced disability, thereby increasing function and improving quality of life in patients experiencing neurological illness or injury. The ArmeoSpring has potential to decrease cost for both the provider and patient over time while providing more engaging, evidence-based therapy.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral upper extremity hemiparesis/hemiplegia
* Upper extremity Fugl-Meyer Assessment Score between 7-60 (Neither hemiplegic nor fully recovered motor function of the shoulder, elbow, wrist)

Exclusion Criteria:

* Inability to follow 1-2 step commands
* Fixed joint contracture
* Unable to tolerate repetitious movement exhibited by pain greater than 5 on Likert Scale
* Any device dependent restrictions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Change in Upper Extremity Fugl Meyer Assessment | Baseline, immediately after intervention, 3 month follow up
  Impairment measure of gross and fine motor upper extremity movements

SECONDARY OUTCOMES:
Patient Satisfaction Survey/Enjoyment Scale | Baseline, immediately after intervention, 3 month follow up
  Self-report of experience with device and supervision; 20 question scale with 0= no satisfaction/enjoyment, 100= extremely satisfied
Box and Blocks Test | Baseline, immediately after intervention, 3 month follow up
  Timed measure of gross manual dexterity
Grip Strength | Baseline, immediately after intervention, 3 month follow up
  Measure of force generated by exerting maximal grip
Short Form Health Survey- 36 | Baseline, immediately after intervention, 3 month follow up
  Self-report questionnaire of health status; minimum score of 0= severe disability and 100 = no disability.
Stroke Impact Scale | Baseline, immediately after intervention, 3 month follow up
  Quality of life measure; Consists of 59 items and assesses 8 domains; Minimum score 0= no recovery, Maximum score 100= full recovery

CONTACTS AND LOCATIONS:
Overall Officials: Tomoko Kitago, MD, Principal Investigator — Burke Medical Research Institute
Locations (1):
- Burke Medical Research Institute, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers at this time.

REFERENCES:
- [Result] Wuennemann MJ, Mackenzie SW, Lane HP, Peltz AR, Ma X, Gerber LM, Edwards DJ, Kitago T. Dose and staffing comparison study of upper limb device-assisted therapy. NeuroRehabilitation. 2020;46(3):287-297. doi: 10.3233/NRE-192993. PMID 32250331